CLINICAL TRIAL: NCT02309151
Title: Direct or Subacute Coronary Angiography in Out-of-hospital Cardiac Arrest - a Prospective, Randomized Study
Brief Title: Direct or Subacute Coronary Angiography in Out-of-hospital Cardiac Arrest
Acronym: DISCO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSC001
Record Dates: First submitted 2014-11-17; First posted 2014-12-05 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Out-of-Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate coronary angiography (Experimental): Immediate coronary angiography for out of hospital cardiac arrest patients with no signs of ST elevation on their first ECG after ROSC
  Interventions: Procedure: Immediate coronary angiography
- Not immediate coronary angiography (No Intervention): Coronary angiography with possible coronary intervention may be performed at the discretion of the interventional cardiologist and should preferably not be performed until three days after the cardiac arrest. This strategy is in accordance with standard practice.

INTERVENTIONS:
Procedure: Immediate coronary angiography — Immediate coronary angiography for out of hospital cardiac arrest patients with no signs of ST elevation on their first ECG after ROSC
  Arms: Immediate coronary angiography

SUMMARY:
The overall aim of this prospective, randomized study is to investigate whether acute coronary angiography (within 120 minutes) with a predefined strategy for revascularization, will improve 30-day survival in patients with out of hospital cardiac arrest with no signs of ST-elevation on ECG after Restoration of Spontaneous Circulation (ROSC). The patients will be randomized to a strategy of immediate coronary angiography within 120 minutes or to a strategy of delayed angiography that may be performed three days after the cardiac arrest.

DETAILED DESCRIPTION:
The study is a prospective randomized open label multicenter study with a registry follow up in which patients with out of hospital cardiac arrest without ST-elevation on their first ECG will be randomized to either a strategy of immediate coronary angiography (treatment group) with possible coronary intervention or a strategy of delayed coronary angiography (control group). The study will include in total 1006 patients with Restoration of Spontaneous Circulation (ROSC). Randomization will be done via a web-based module after ECG is taken at the first medical contact but no later than after arrival at the emergency room. Coronary angiography should be performed within 120 minutes from randomization in the immediate angiography group. In the delayed angiography group, angiography with possible coronary intervention will be performed at the discretion of the interventional cardiologist and should preferably not be performed until three days after the cardiac arrest. This strategy is in accordance with standard practice. In case of recurrent chest pain, ST elevation, circulatory instability or cardiogenic shock, cross over to early angiography may occur. The quality of life and health economics will be evaluated at 6 months. The patients will undergo extensive neurocognitive tests and health instruments, these will be analyzed and presented.

ELIGIBILITY:
Inclusion Criteria:

* Witnessed out of hospital cardiac arrest
* Restoration of Spontaneous Circulation (ROSC) >20 minutes
* Coronary angiography is expected to be performed within 120 minutes from inclusion and randomization at hospital

Exclusion Criteria:

* Patient age <18 years
* Obvious extracardiac genesis of cardiac arrest such as trauma, hemorrhagic shock, and / or asphyxia (eg drowning, suffocation, hanging, exposure to fire smoke)
* Terminally ill patients with a life expectancy of less than 1 year
* Patients with ST-elevation
* Known pregnancy
* Patient awake GCS >8 (Glasgow Coma Scale)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1006 (Estimated)
Dates: Start 2014-12; Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
30 day survival | 30 days
  Follow up will be performed at 30 days, telephone call or visit.

SECONDARY OUTCOMES:
Survival with good neurological function | 30 days
  30-day survival and a follow up of health status, functional outcome associated to cerebral performance and general functional outcome/activities of daily living
Survival at discharge from ICU (individual for each subject) and at 6-months | At discharge from ICU, an expected average of 3-30 days and at 6-months
  Recorded in the e-CRF (electronic Case Report Form)
Survival with good neurological function at discharge from ICU and 6-months | At discharge from ICU, an expected average of 3-30 days and at 6-months
  Survival with good neurological function at discharge and at 6-months. Assessing functional outcome associated to cerebral performance and general functional outcome/activities of daily living and also global functional outcome, independent living and social reintegration at 6-months
Cardiac function | 72 hours and at 6 months
  Measured with echocardiography
Follow up of neurological function at 6-months | Measured at 6 months
  A 6 month follow up of neurological function will be assessed by validated screening battery in OHCA (Out of Hospital Cardiac Arrest) patients in general functional outcome, activities of daily living, cognitive functioning, attention, anxiety and depression, fatigue, cardiac disease specific health and care giver burden.
Hemodynamic parameters (urine output, highest lactate and vasopressor/inotropic support) | During ICU care (maximum of 7 days)
  Parameters measured daily during ICU care
ECG findings compared to findings at coronary angiography | During hospital stay up to a maximum of 6-months
  Primary ECG, performed in the pre-hospital setting or at the emergency department, will be compared with findings at coronary angiography intervention (performed immediately or later during hospital stay depending on randomisation)

CONTACTS AND LOCATIONS:
Overall Officials: Sten Rubertsson, Md,PhD, Principal Investigator — Uppsala Universtiy hospital
Locations (21):
- Denmark (3):
  - Aalborg University hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Odense University hospital, Odense
- Netherlands (8):
  - Amsterdam UMC, Amsterdam
  - Albert Schweitzer Hospital, Dordrecht
  - Catharina Ziekenhuis, Eindhoven
  - Treant Hospital, Emmen
  - Zuyderland Hospital, Heerlen
  - Antonius Hospital, Nieuwegein
  - Radboud University Medical Center, Nijmegen
  - Haaglanden Medisch Centrum, The Hague
- Sweden (10):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Karolinska Universitetssjukhuset, Huddinge
  - Skånes Universitetssjukhus, Lund
  - Skåne Universitetssjukhus, Malmo
  - Örebro Universitetssjukhus, Örebro
  - Karolinska Universitetssjukhuset, Solna
  - Danderyd Sjukhus, Stockholm
  - Södersjukhuset AB, Stockholm
  - Umeå Universitetssjukhus, Umeå
  - Uppsala University hospital, Uppsala

REFERENCES:
- [Derived] Elfwen L, Lagedal R, Rubertsson S, James S, Oldgren J, Olsson J, Hollenberg J, Jensen U, Ringh M, Svensson L, Nordberg P. Post-resuscitation myocardial dysfunction in out-of-hospital cardiac arrest patients randomized to immediate coronary angiography versus standard of care. Int J Cardiol Heart Vasc. 2020 Mar 2;27:100483. doi: 10.1016/j.ijcha.2020.100483. eCollection 2020 Apr. PMID 32154359
- [Derived] Elfwen L, Lagedal R, Nordberg P, James S, Oldgren J, Bohm F, Lundgren P, Rylander C, van der Linden J, Hollenberg J, Erlinge D, Cronberg T, Jensen U, Friberg H, Lilja G, Larsson IM, Wallin E, Rubertsson S, Svensson L. Direct or subacute coronary angiography in out-of-hospital cardiac arrest (DISCO)-An initial pilot-study of a randomized clinical trial. Resuscitation. 2019 Jun;139:253-261. doi: 10.1016/j.resuscitation.2019.04.027. Epub 2019 Apr 24. PMID 31028826
- [Derived] Lagedal R, Elfwen L, James S, Oldgren J, Erlinge D, Ostlund O, Wallin E, Larsson IM, Lilja G, Cronberg T, Rubertsson S, Nordberg P. Design of DISCO-Direct or Subacute Coronary Angiography in Out-of-Hospital Cardiac Arrest study. Am Heart J. 2018 Mar;197:53-61. doi: 10.1016/j.ahj.2017.11.009. Epub 2017 Dec 5. PMID 29447784